CLINICAL TRIAL: NCT00003129
Title: Phase II Study of Intravesical Therapy With AD 32 in Patients With Papillary Urothelial Carcinoma or Carcinoma in Situ (CIS) Refractory to Prior Therapy With Bacillus Calmette-Guerin
Brief Title: Chemotherapy in Treating Patients With Early-Stage Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065892; E-3897
Record Dates: First submitted 1999-11-01; First posted 2003-04-18 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — valrubicin

INTERVENTIONS:
Drug: valrubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy in treating patients with early-stage bladder cancer that has not responded to BCG therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recurrence rate and disease free survival in patients with recurrent or refractory papillary transitional cell carcinoma of the bladder with or without carcinoma in situ of the bladder treated with intravesical AD 32.
* Evaluate the safety of administering this drug in these patients.
* Determine the effectiveness of this drug, in terms of recurrence rates and disease free survival, in these patients.

OUTLINE: Patients are stratified according to cellular diagnosis (papillary transitional cell carcinoma (Ta/T1) with no carcinoma in situ (Tis) vs Tis with or without Ta/T1).

Patients receive intravesical AD 32 once a week for 6 weeks.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent superficial bladder cancer defined as papillary transitional cell carcinoma (stage Ta/T1) and/or carcinoma in situ (stage Tis) of the urinary bladder

  * No evidence of invasion of the underlying muscle (stage T2) at baseline
* Must meet 1 of the following criteria:

  * Failure of at least 2 prior courses of intravesical therapy, 1 of which must have been a course of BCG
  * Recurrent or persistent disease within 6 months after failing a 6-week course of BCG followed by maintenance therapy
  * Inability or ineligibility to complete 1 course of intravesical therapy with BCG, and failure of 2 prior courses of intravesical therapy with an alternative agent
* Diagnosis must have been made no more than 24 months after completion of prior treatment with intravesical immunotherapy or chemotherapy
* If carcinoma in situ is current or previous diagnosis, the biopsies must be obtained from at least 4 sites (bladder mapping)
* If prostatic urothelial biopsy discloses carcinoma in situ, transurethral prostatic resection must be carried out prior to study
* Papillary disease must have undergone complete transurethral resection (TURBT) within 28 days before study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT and SGPT less than 3 times ULN

Renal:

* Creatinine no greater than 2.5 mg/dL

Other:

* Normal upper tract (ureter and renal pelvic) evaluation within 6 months
* No known sensitivity to anthracyclines or to Cremophor EL
* HIV negative
* No known AIDS or HIV-1 associated complex
* No other significant concurrent illness
* No other prior malignancy within the past 3 years except superficial bladder cancer, adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent biological response modifier therapy

Chemotherapy:

* See Disease Characteristics
* Prior oral bropirimine for bladder cancer allowed
* No prior AD 32 for bladder cancer
* No other intravenously administered systemic chemotherapy for bladder cancer
* No concurrent chemotherapy for any other malignancy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* No prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 1998-09-01 (Actual); Primary Completion 2002-11 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Ignatoff, MD, Study Chair — Endeavor Health
Locations (10):
- United States (10):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin

REFERENCES:
- [Result] Ignatoff JM, Chen YH, Greenberg RE, Pow-Sang JM, Messing EM, Wilding G. Phase II study of intravesical therapy with AD32 in patients with papillary urothelial carcinoma or carcinoma in situ (CIS) refractory to prior therapy with bacillus Calmette-Guerin (E3897): a trial of the Eastern Cooperative Oncology Group. Urol Oncol. 2009 Sep-Oct;27(5):496-501. doi: 10.1016/j.urolonc.2008.05.004. Epub 2008 Jul 17. PMID 18639470